CLINICAL TRIAL: NCT01194934
Title: A Single Center, Open-label, Repeated Dose, Phase I Study in Healthy Subjects to Assess the Safety, Tolerability, Pharmacokinetics and the Effect on Mobilization of Hematopoietic Stem Cells of NOX-A12 Alone and in Combination With Filgrastim
Brief Title: NOX-A12 Multiple Ascending Dose Study in Healthy Volunteers
Acronym: SNOXA12C101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TME Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNOXA12C101; 2010-020937-14 (EudraCT Number)
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Stem Cell Transplantation; SDF-1; L-oligonucleotide Aptamer; Spiegelmer; Hematopoietic Stem Cells
MeSH Terms: interventions — NOX-A12; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Experimental): Group A: 2.0 mg/kg NOX-A12 IV every day for 5 days
  Interventions: Drug: NOX-A12
- Group B (Experimental): Group B: 4.0 mg/kg NOX-A12 IV every day for 5 days
  Interventions: Drug: NOX-A12
- Group C (Active Comparator): The treatment groups will enter the study sequentially. The decision on starting groups C and D will be made after groups A and B have been completed and data are available.
  Group C: 5 µg/kg filgrastim SC every day for 5 days
  Interventions: Drug: Filgrastim
- Group D (Experimental): The treatment groups will enter the study sequentially. The decision on starting groups C and D will be made after groups A and B have been completed and data are available.
  Group D: Safe and efficacious dose of NOX-A12 IV in combination with filgrastim SC for 5 days
  Interventions: Drug: NOX-A12 in combination with Filgrastim

INTERVENTIONS:
Drug: NOX-A12 — 4 mg/kg daily IV for 5 days
  Other Names: olaptesed pegol
  Arms: Group B
Drug: NOX-A12 — 2 mg/kg daily IV for 5 days
  Other Names: olaptesed pegol
  Arms: Group A
Drug: Filgrastim — 5 µg/kg SC daily for 5 days
  Other Names: olaptesed pegol
  Arms: Group C
Drug: NOX-A12 in combination with Filgrastim — Safe and efficacious dose regimen according to results of groups A and B
  Other Names: olaptesed pegol
  Arms: Group D

SUMMARY:
This is the second clinical study of NOX-A12. This study intends to provide information on the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of repeated intravenous doses of NOX-A12 (2.0 and 4.0 mg/kg/d) alone and to compare the mobilization of hematopoietic stem cells (HSC) obtained with NOX-A12 alone with that obtained in combination with filgrastim in healthy subjects. A single center, open-label, repeated dose study design is selected to best address the study objectives.The results from this study will establish the basis for further development of NOX-A12 in lymphoma patients undergoing autologous hematopoietic stem cell transplantation

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed by the subject.
2. Healthy male and female subjects aged 18 to 55 years of any ethnic origin.
3. Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, laboratory tests and ECG. Values out of reference range have to be assessed as not clinically significant (NCS) or clinically significant (CS) by the investigator. Individuals presenting deviating values assessed as not clinically significant may be included.
4. Male subjects willing to use contraceptive methods from the time of dosing until 3 months after study drug administration (such as condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository), females must be of non-childbearing potential. Non-childbearing potential is defined as follows: Female subjects must be surgically sterile or post-menopausal (defined as at least two years post cessation of menses and follicular stimulating hormone ≥ 35 mIU/mL and serum estradiol ≤25 pg/mL), non-lactating and have a negative pregnancy test.
5. Body mass index between 19 and 29 kg/m2 (extremes included).
6. Body weight between 50 and 100 kg (extremes included).
7. Calculated creatinine clearance ≥ 90 mL/min according to the Cockcroft-Gault-formula.
8. Normal lung function (FVC and FEV1 at least 80% of predicted values) at screening.
9. O2 saturation between 96% and 100% (extremes included) at screening.
10. The subject is co-operative and available for the entire study.

Exclusion Criteria:

1. Evidence in the subject's medical history or in the medical examination of any clinically significant hepatic, renal, gastrointestinal, cardiovascular, pulmonary, hematological or other significant acute or chronic abnormalities which might influence either the safety of the subject or the absorption, distribution, metabolism or excretion of the active agent under investigation.
2. History of general malignant diseases.
3. History of renal calculus.
4. Hypersensitivity to drugs, atopic eczema, allergic bronchial asthma or any clinically significant allergic disease (excluding non-active hayfever).
5. Hypersensitivity to the active substances or to any of its excipients.
6. Subjects having already received G-CSF in the past.
7. Intake of vitamin A derivates or retinoids within 30 days prior to the start of study drug administration.
8. Subjects who have a significant history of sensitivity to natural sunlight or artificial light such as ultraviolet (UV) light from sunbeds.
9. History of thrombosis or increased bleeding risk.
10. Laboratory test results outside the reference values as laid down by the study center, which may be an evidence of disease. Positive result of HIV1/2, HCV antibody or HBs antigen testing.
11. Subjects who have an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risk of participating in the study, such as QTcB interval >450 msec (females) and >430 msec (males), 2nd or 3rd degree atrioventricular block, complete left bundle branch block, complete right bundle branch block or Wolff-Parkinson-White Syndrome, defined as PR<110 msec, confirmed by a repeated ECG.
12. Subjects who have had a clinically significant illness within 8 weeks prior to the start of study drug administration as determined by the investigator.
13. History of relevant heart disorders or evidence of hyper- or hypotension (supine blood pressure systolic >140 mmHg or <95 mmHg or diastolic >90 mmHg or <65 mmHg at screening).
14. Bradycardia or bradyarrhythmia (heart rate after 3 minutes supine rest <45/min at screening).
15. Tachycardia or Tachyarrhythmia (heart rate after 3 minutes supine rest >90/min at screening).
16. Chronic infection or acute infection or fever within the last 8 weeks prior to the start of study drug administration as determined by the investigator.
17. Subjects who have received any prescribed systemic or topical medication within 14 days prior to dose administration as stated by the subject at screening, unless the medication will not interfere with the study procedures or compromise safety as assessed by an investigator in consultation with the sponsor.
18. Subjects who have received any medications (including St John's Wort) known to chronically alter drug absorption or elimination processes within 30 days prior to study drug administration as stated by the subject at screening, unless the medication will not interfere with the study procedures or compromise safety as assessed by an investigator in consultation with the sponsor.
19. Single use of any medication (including OTC) that are not expressively permitted within two weeks prior to scheduled admission to the study (self-medication or prescription) as stated by the subject at screening, unless the medication will not interfere with the study procedures or compromise safety as assessed by an investigator in consultation with the sponsor.
20. Abuse of alcohol (equivalent to more than 18 units per week, where 1 unit is equivalent to one beer (about 330 ml) or one wine (about 150 ml) or one drink (about 40 ml)), caffeine (equivalent to more than 750 mg per day) or tobacco (equivalent to more than 10 cigarettes a day).
21. Alcohol breath test positive at screening.
22. Drug addiction, positive drug screening in urine.
23. Participation in another clinical investigation or being in the restriction period after a clinical investigation.
24. Blood donation of more than 100 ml or a comparable blood loss within three months prior to study drug administration.
25. Subjects who are known or suspected (i) not to comply with the study directives, (ii) not to be reliable or trustworthy, (iii) not to be capable of understanding and evaluating the information given to them as part of the formal information policy (informed consent), in particular regarding the risks and discomfort to which they would agree to be exposed to, or (iv) to be in such a precarious financial situation that they no longer weigh up the possible risks of their participation and the unpleasantness they may be involved in.
26. Subjects with inadequate venous access.
27. Subjects who, in the opinion of the investigator, should not participate in the study.
28. Subjects with an abnormal splenic size.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of repeated doses of NOX-A12 alone and in combination with filgrastim in healthy subjects. | 1 month

SECONDARY OUTCOMES:
To determine the pharmacokinetics of repeated doses of NOX-A12 alone and in combination with filgrastim in healthy subjects. | 1 month
To quantify the mobilization of HSCs in peripheral blood after repeated doses of NOX-A12 alone, of filgrastim alone and after the combination of NOX-A12 with filgrastim. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Frank Fliegert, MD, Study Director — TME Pharma AG
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany